CLINICAL TRIAL: NCT03530098
Title: Prospective, Multi-Center, Randomized Controlled Trial for Skeletal Age Assessment AI Model
Brief Title: Validation of an Artificial Intelligence-based Algorithm for Skeletal Age Assessment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Safwan S Halabi, MD, Principal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB #44764
Record Dates: First submitted 2018-05-07; First posted 2018-05-21 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Bone Age
Keywords: Age Determination by Skeleton; Machine Learning; Deep Learning; Artificial Intelligence; Prospective; Clinical Validation

STUDY DESIGN:
Intervention Model Description: A hand radiograph will be randomly assigned to one of two groups - control and experiment. In the control group, participating radiologists will diagnose the exam using the current standard of care (no intervention). In the experiment group, the radiologists will factor in the output of the Artificial Intelligence algorithm in their skeletal age estimation. In all cases, the decision of the radiologist will be considered final.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Control (Without-AI) (No Intervention): This is the control arm where no intervention is provided; represents current standard of care.
- Experiment (With-AI) (Experimental): This is the experiment arm where the intervention, "BoneAgeModel", is provided. The participating radiologists in this arm will receive the output of the Artificial Intelligence algorithm. They will be asked to incorporate this new information with their normal workflows to make a diagnosis. The radiologists' diagnosis will be considered final.
  Interventions: Device: BoneAgeModel

INTERVENTIONS:
Device: BoneAgeModel — BoneAgeModel is an Artificial Intelligence tool that takes in a hand radiograph and gender, and outputs the skeletal (bone) age. The intervention involves using this tool as a factor in the clinical decision making process of the participating radiologists. The radiologist's decision will be considered final.
  Arms: Experiment (With-AI)

SUMMARY:
The purpose of this study is to understand the effects of using an Artificial Intelligence algorithm for skeletal age estimation as a computer-aided diagnosis (CADx) system. In this prospective real-time study, the investigators will send de-identified hand radiographs to the Artificial Intelligence algorithm and surface the output of this algorithm to the radiologist, who will incorporate this information with their normal workflows to make an estimation of the bone age. All radiologists involved in the study will be trained to recognize the surfaced prediction to be the output of the Artificial Intelligence algorithm. The radiologists' diagnosis will be final and considered independent to the output of the algorithm.

DETAILED DESCRIPTION:
The investigators are targeting to study the effect of their Artificial Intelligence algorithm on the radiologists' estimation of skeletal age. Currently, radiologists make the estimation using only the radiographic images and health records. As part of this study, the radiologists will estimate skeletal age from radiographic images, health records, and the output of the CADx algorithm. The investigators wish to understand how radiologists using the Artificial Intelligence algorithm compare to radiologists who do not for the specific task of estimating skeletal age.

This study is organized as a multi-institutional randomized control trial with two arms - experiment (receiving the Artificial Intelligence algorithm's output) and control (no intervention). Both of these arms will be compared to a clinical reference standard ("gold standard") composed of a panel of radiologists. The metric of comparison will be Mean Absolute Distance (MAD). The investigators plan to use statistical tests such as the t-test to determine any statistically-significant difference in skeletal age estimation between the two groups.

The investigators have recruited and analyzed data from a sample size of 1600 exams. Patients getting these exams will not undergo any research procedures that deviate from the current standard practices.

ELIGIBILITY:
Exams that meet the following inclusion criteria will be included: (1) exams read by radiologists who interpret pediatric skeletal age exams and verbally consent to participate (2) exams that contain a procedure code or study description indicative of a skeletal age exam.

Exams containing more than one radiograph will not be included. Exams for which a trainee provides a preliminary interpretation will be excluded. No further exclusion criteria will be applied on the basis of image quality metrics or manufacturers. No exclusion criteria will be applied on the basis of patient chronological age.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1903 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Langlotz, M.D. Ph.D., Study Chair — Stanford University; David Eng, B.S., Study Director — Stanford University; Nishith Khandwala, B.S., Study Director — Stanford University; Safwan Halabi, M.D., Principal Investigator — Stanford University
Locations (6):
- United States (6):
  - Stanford University, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Boston Children's Hospital, Boston, Massachusetts
  - New York University, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

RESULTS

PARTICIPANT FLOW:
Groups:
- Control (Without-AI): Diagnosis by radiologists made according to current standard of care methods.
- Experiment (With-AI): Diagnosis by radiologists informed by "BoneAgeModel" Artificial Intelligence (AI) algorithm incorporated into normal radiologist workflows and considered as a factor in the clinical decision making process. The radiologists' diagnosis will be considered final. BoneAgeModel takes in a hand radiograph and gender, and outputs the skeletal (bone) age.
Period: Overall Study
Arm/Group | Control (Without-AI) | Experiment (With-AI)
Started | 939 | 964
Ground-truth Labeled (Ground-truth labeled: exam was interpreted by a panel of 4 radiologists and their interpretations were averaged to determine a final label.) | 741 | 794
Primary Analysis Set (Primary analysis set: Participants with ground-truth labeled exam results and no bone deformity.) | 739 | 792
Completed | 939 | 964
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Primary analysis set: Participants with ground-truth labeled exam results and no bone deformity.
  Ground-truth labeled: exam was interpreted by a panel of 4 radiologists and their interpretations were averaged to determine a final label.
Groups:
- Experiment (With-AI): Diagnosis by radiologists informed by "BoneAgeModel" AI algorithm incorporated into normal radiologist workflows and considered as a factor in the clinical decision making process.
- Total: Total of all reporting groups
Arm/Group | Control (Without-AI) | Experiment (With-AI) | Total
Number analyzed (Participants) | 739 | 792 | 1531
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.8 (3.6) | 11.5 (3.6) | 11.7 (3.6)
Age, Customized [Count of Participants; unit: Participants]
  0-4 years | 12 | 14 | 26
  >4-8 years | 110 | 131 | 241
  >8-12 years | 206 | 249 | 455
  >12-16 years | 331 | 338 | 669
  >16-20 years | 75 | 57 | 132
  >20 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 338 | 359 | 697
  Male | 401 | 433 | 834
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 739 | 792 | 1531
Skeletal age final impression (mean) [Mean (Standard Deviation); unit: years] — Final impression is the baseline radiologist assessment.
  years | 11.6 (3.6) | 11.4 (3.5) | 11.5 (3.5)
Skeletal age final impression (categorical) [Count of Participants; unit: Participants] — Final impression is the baseline radiologist assessment.
  Participants
    0-4 years | 21 | 17 | 38
    >4-8 years | 110 | 131 | 241
    >8-12 years | 191 | 223 | 414
    >12-16 years | 344 | 362 | 706
    >16-20 years | 73 | 59 | 132
    >20 years | 0 | 0 | 0
Clinical histories [Count of Participants; unit: Participants] — Clinical history types
  Participants
    Endocrine | 391 | 430 | 821
    Orthopedic | 82 | 63 | 145
    Congenital/syndrome | 9 | 12 | 21
    Medical | 16 | 17 | 33
    Other | 4 | 12 | 16
    More than one category | 20 | 17 | 37
    Not available | 217 | 241 | 458

OUTCOME MEASURES:

1. Primary Outcome: Paired Difference of Skeletal Age Estimate
Description: Mean absolute difference between dictated final impressions (baseline measure by Radiologist) and the consensus determination of a panel of radiologists following review.
Time Frame: Up to 10 minutes to acquire the scan; up to 2 days to complete diagnosis review
Population: as for baseline characteristics
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Control (Without-AI) | Experiment (With-AI)
Number analyzed (Participants) | 739 | 792
months | 5.95 [5.53 to 6.37] | 5.36 [5.01 to 5.71]
Statistical Analysis 1: Comparison: Control (Without-AI) vs Experiment (With-AI); Test type: Superiority; p = 0.04, t-test, 2 sided; Odds Ratio (OR) = -0.59, 95% CI 2-sided [-1.14 to -0.04]

2. Secondary Outcome: Time for Diagnosis
Description: Amount of time taken by radiologists when using the BoneAgeModel as compared to when they are not.
Time Frame: Up to approximately 4 minutes
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Experiment (Without-AI): Diagnosis by radiologists informed by "BoneAgeModel" AI algorithm incorporated into normal radiologist workflows and considered as a factor in the clinical decision making process.
Arm/Group | Control (Without-AI) | Experiment (Without-AI)
Number analyzed (Participants) | 739 | 792
seconds | 142 [80 to 248] | 102 [59 to 196]
Statistical Analysis 1: Comparison: Control (Without-AI) vs Experiment (Without-AI); Test type: Other; p = 0.001, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: Day of study visit (average approximately 1 hour)
Arm/Group | Control (Without-AI) | Experiment (With-AI)
All-Cause Mortality (participants affected / at risk) | 0/939 | 0/964
Serious Adverse Events (participants affected / at risk) | 0/939 | 0/964
Other Adverse Events (participants affected / at risk) | 0/939 | 0/964

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT03530098/Prot_SAP_000.pdf